CLINICAL TRIAL: NCT01106768
Title: Evaluation of Oral Needs of Children With Disorder Attention Deficit/Hyperactivity Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-A00616-49
Record Dates: First submitted 2010-04-09; First posted 2010-04-20 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: oral health needs; children; attention deficit disorder with or without hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- test cohort: Evaluation of oral health needs of children with attention deficit disorder with or without hyperactivity
- not disorder cohort: children without attention deficit disorder

SUMMARY:
There is little accurate data in the literature at present on oral problems of hyperactive children, especially regarding care needs that would justify an assumption oral specific. The purpose of this study is therefore to have accurate data regarding the risk of caries, other oral diseases like periodontal disease, trauma, and assess the needs dental care and problems in cooperation for dental care in a population of children and adolescents with hyperactivity disorder with attention deficit. Finally, it has recently been described as the sleep disordered breathing was not uncommon in disorder attention deficit/hyperactivity disorder, whether snoring and/or apnea. But it is now accepted that some features of facial morphology favoring pharyngeal congestion occur in individuals with obstructive sleep apnea (hyperdivergent typology with increased anterior facial height and decreased posterior facial height, becoming the facial retrognathia, pharyngeal congestion, elongation and thickening of the soft palate, low position of the hyoid bone). A cephalometric analysis of craniofacial architecture and relationships with the soft tissue surrounding skeletal structures will detect if any of these specific characteristics that could promote sleep disordered breathing are found in disorder attention deficit/hyperactivity disorder prevalence with a particular.

ELIGIBILITY:
Inclusion Criteria:

* Consent signed by parents before the examination
* With of a social security scheme
* Age greater than or equal to 5 years and less than 15 years, Children with a diagnosis of attention deficit / hyperactivity confirmed or made by a physician specialists co-investigators of the study, diagnosis defined according to precise criteria for a disorder attention deficit/hyperactivity disorder as specified in DSM-IV with a normal IQ, ie higher than 80, and without other neurological or psychiatric
* Child consultant in a hospital or doctors' offices

Exclusion Criteria:

* Refusal of consent of the parents
* No affiliation to a social security scheme
* Age below 5 years or more than 15 years
* Diagnosis of a disorder attention deficit/hyperactivity disorder not confirmed by a physician , IQ <80, Pathology associated neurological or psychiatric

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children with attention deficit disorder with or without hyperactivity
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2009-05; Primary Completion 2013-04 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Cod and CAOD index for caries,PI and GI indices for periodontal disease, dysfunction and malocclusion classification by WHO and Analysis cephalometric | 18 months

SECONDARY OUTCOMES:
Measurement of anxiety through the CFSS-DS scale (Dental subscale of Children's Fear Survey Schedule, Schedule 1) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: MANIERE Marie-Cécile, MD, Principal Investigator — not affiliated
Locations (1):
- CHRU ,Hopital Civil, Département d'Odontologie Pédiatrique Service de Consultations et de Traitements Dentaires, Strasbourg, France